CLINICAL TRIAL: NCT02699216
Title: BioCurrent Electrical Stimulation for the Treatment of Dry Age-Related Macular Degeneration
Brief Title: BioCurrent Electrical Stimulation for the Treatment of Dry ARMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: DuBois Vision Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WSW001
Record Dates: First submitted 2016-02-16; First posted 2016-03-04 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Dry Macular Degeneration
Keywords: Macular Degeneration; Eye Diseases; Retinal Degeneration; Retinal Diseases
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Eye Diseases; Retinal Degeneration; Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 Active Treatment (Experimental): Subjects will undergo 8 treatments, approximately 11 minutes, to the enrolled eyes daily for three consecutive days, with an active device. They will receive no treatments on day 4 and 5.
  Interventions: Device: Electrical Stimulation of the Retina
- Phase 1 Sham Treatment (Placebo Comparator): Subjects will undergo 8 sham treatments, approximately 11 minutes, with a non-functional device to the enrolled eyes daily for three consecutive days during week 1, with no treatments on day 4 and 5. Followed by 8 active treatments, for approximately 11 minutes, for three consecutive days, with an active device during week 2, with no treatments on day 4 and 5.
  Interventions: Device: Electrical Stimulation of the Retina
- Phase 2 Open Label (Experimental): Subjects will undergo 8 treatments, approximately 11 minutes, to the enrolled eyes daily for three consecutive days, with an active device. They will receive no treatments on day 4 and 5.
  Interventions: Device: Electrical Stimulation of the Retina

INTERVENTIONS:
Device: Electrical Stimulation of the Retina — Transpalpebral micro-current electrical stimulation treatment for 3 consecutive days followed by a short wash-out period of 2 days.

SUMMARY:
This study evaluates the treatment of Dry Macular Degeneration and the resulting change in vision with a very, very low current that is similar to what occurs in the body naturally. In Phase 1, 16 participants will be treated, with half receiving treatment and half a sham (no treatment). After the treatment period of one week, those not treated will be treated. In Phase 2, all participants will be treated.

DETAILED DESCRIPTION:
The study will assess the effectiveness of transpalpebral micro-current electrical stimulation on improving the visual acuity in subjects with vision loss from Dry Macular Degeneration. The BioCurrent electrical stimulation will be applied by a device with the intended use of treating Dry Macular Degeneration. The device delivers a micro-current, an electrical current in the one millionth of an ampere range, to the retina in frequencies changing in a pre-defined pattern from 5Hz to 80Hz during each spot (40 sec). The device also incorporates a voltage limiter (a maximum of 245 micro A is possible) and a current level indicator. 200 micro A will be used. Very low electrical micro-current is delivered to the subject through the goggle probe.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity can be no better than 20/40 and no worse than 20/200 for each enrolled eye
* Confirmed diagnosis of Dry MD
* Vision loss attributable to Dry MD
* Subjects must be highly motivated, alert, oriented, mentally competent and able to understand and comply with the requirements of the study, abide by the restrictions, return for all required visits, and provide voluntary informed consent

Exclusion Criteria:

* Any retinal pathology other than Dry MD
* Evidence or history of wet MD
* Previous intravitreal injection
* Seizure disorders
* Dense cataract
* Eyelid pathology at the treatment sites
* Any prior electrical micro-stimulation treatment to the eyes
* Poor general health
* Active cancer
* Life expectancy less than 12 months
* Non-ambulatory
* Not considered suitable for participation for any other reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Best-corrected Visual Acuity using the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart | Baseline, Day 5
  Significant changes in ETDRS visual acuity; baseline and Day 5.

SECONDARY OUTCOMES:
Changes in retinal sensitivity assessed by Microperimetry | Baseline, Day 5
  Significant Changes in retinal sensitivity; baseline and Day 5.

IPD SHARING:
Plan to Share IPD: No